CLINICAL TRIAL: NCT06624605
Title: Enhancing Interdisciplinary Understanding of Ophthalmology Notes Through Local Large Language Model
Brief Title: Enhancing Interdisciplinary Understanding of Ophthalmology Notes Through a Local Large Language Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John J Chen (Other)
Responsible Party: Sponsor-Investigator, John J Chen, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-000550
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Communication; Artificial Intelligence (AI); Artificial Intelligence Technology; Interdisciplinary Communication
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: Randomized study assessing the efficacy of Large Language Model-generated Plain Language Summaries of Ophthalmology notes in increasing non-ophthalmologist note understanding. Notes were randomized to intervention (Summary + Original Note) or control (Original note only) arms. Non-ophthalmology providers were sent surveys assessing note comprehension for both control and treatment arm notes, and Ophthalmologists were sent surveys for intervention arm notes regarding Summary accuracy and other attributes. Conducted as a Quality Improvement initiative.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants receive standard ophthalmology notes without any additions.
- Intervention (Experimental): Participants receive standard ophthalmology notes with an appended LLM-generated plain language summary, reviewed and edited by the ophthalmologist. The plain language summary is clearly marked as generated as part of a Quality Improvement initiative.
  Interventions: Other: Large Language Model-generated Plain Language Summary of Ophthalmology notes

INTERVENTIONS:
Other: Large Language Model-generated Plain Language Summary of Ophthalmology notes — Prospective, randomized Quality Improvement study with real-world implementation of Large Language Model-generated Plain Language Summaries of Ophthalmology notes.
  Arms: Intervention

SUMMARY:
This prospective, randomized controlled trial evaluated the efficacy of adding Large Language model (LLM)-generated Plain Language Summaries (PLSs) to Standard Ophthalmology Notes (SONs) in enhancing comprehension among non-ophthalmology providers. The study utilized surveys to assess non-ophthalmology providers' comprehension and satisfaction with the notes and ophthalmologists' evaluation of PLS accuracy, safety, and time burden. An objective semantic and linguistic analysis of the PLSs was also conducted.

ELIGIBILITY:
Inclusion Criteria:

* Evaluation by an Ophthalmologist in the Mayo Clinic Department of Ophthalmology in Rochester, MN in either the inpatient or outpatient setting between Feb 1, 2024 - May 31, 2024.

Exclusion Criteria:

* No in-network non-Ophthalmologist care providers in the medical record
* Procedure-only visits containing only a procedure note

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Non-Ophthalmologist Note Comprehension and Satisfaction | From enrollment to 8 weeks after enrollment
  Assessed via survey responses evaluating understanding of the patient&amp;#39;s ophthalmology diagnosis, satisfaction with the note, and overall preference between Standard Ophthalmology Note and Standard Ophthalmology Note + Plain Language Summary.
  Degree of understanding was assessed on the following Likert scale:
  Not at all Neutral Moderately A great deal
  Satisfaction was graded on the following Likert scale:
  Not satisfied at all Somewhat unsatisfied Neutral Somewhat satisfied Satisfied
  Preference between note types was assessed on the following Likert scale:
  Standard Note, a great deal Standard Note, somewhat Neutral Plain Language Summary, somewhat Plain Language Summary, a great deal

SECONDARY OUTCOMES:
Ophthalmologist Evaluation of Summary Accuracy and Time burden | Assessed at a single time point <24 hr after enrollment
  Assessed via survey responses regarding Plain Language Summary accuracy in reflecting the Standard Ophthalmology Note findings, time spent reviewing/editing, and perceived burden.
  Accuracy in reflecting findings was graded on the following Likert scale:
  Not at all Neutral A little A great deal
  Time spent reviewing/editing was reported using the following options:
  <1 minute
  1. minute
  2. minutes
  3. minutes
  4. minutes
  5. or more minutes
  Perceived burden was graded on the following Likert scale:
  Not at all Neutral A little A great deal
Semantic and Linguistic Quality of Plain Language Summaries | Assessed at a single time point <24 hr following enrollment
  Flesch Reading Ease
  Scale: 0 (poor) to 100 (good)
Semantic and Linguistic Quality of Plain Language Summaries | Assessed at a single time point <24 hr following enrollment
  Flesch-Kincaid Grade Level
  Scale: 0 (most difficult to read, highest grade level) to 80 (easiest to read, lowest grade level)
Semantic and Linguistic Quality of Plain Language Summaries | Assessed at a single time point <24 hr following enrollment
  Semantic Measure of Gobbledygook (SMOG) Index
  Scale: 0 (easiest to read) to 11 (most difficult to read)
Semantic and Linguistic Quality of Plain Language Summaries | Assessed at a single time point <24 hr following enrollment
  BERTScore Measure of Linguistic Similarity
  Scale: -1 (least similar) to +1 (most similar)
Semantic and Linguistic Quality of Plain Language Summaries | Assessed at a single time point <24 hr following enrollment
  SBERT Cosine Similarity Measure of Linguistic Similarity
  Scale: -1 (least similar) to +1 (most similar)

OTHER OUTCOMES:
Presence of Errors, Type of Errors, and Potential Harm of Errors | Assessed at a single time point &amp;amp;lt;24 hr following enrollment and again at a single time point 8 weeks after enrollment
  Presence of any incorrect or missing information in the Plain Language Summary, error rates, types of errors, and potential harm rating.
  Types of errors were reported as:
  HPI Exam findings Diagnosis Plan Explanation of the patient's overall eye health Other N/A
  Likelihood of harm was graded on the following scale:
  Low risk Medium risk High risk N/A
  Potential harm rating was graded on the following scale:
  Mild or moderate harm Death or severe harm

CONTACTS AND LOCATIONS:
Overall Officials: John J Chen, MD, PhD, Study Director — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Beginning after publication with no end date
Access Criteria: The underlying data supporting the findings of this study can be made available to clinical investigators and researchers upon request. Written requests for data sharing including an analysis plan will be required before approval. These requests will be individually assessed in consultation with the study team leads and co-investigators as appropriate. If other investigators are interested in performing additional analyses, these requests can be made to the corresponding author (PDT) and analyses will be performed in collaboration with the Mayo Clinic. In all cases, any data and materials to be shared will be released via a Material Transfer Agreement. Individual-level data will be available and data sharing will ensure that the rights and privacy of individuals participating in the research always remains protected. The anticipated time frame to respond to initial data requests is 1 month.